CLINICAL TRIAL: NCT07255261
Title: Post-Marketing Clinical Follow Up On Hyaluronic Acid-Based Dermal Fillers Using COLD-X™ Technology By Symatese
Brief Title: Evaluation of Facial HA Dermal Fillers in Real-Life Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Symatese (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN2108_CIP
Record Dates: First submitted 2025-11-14; First posted 2025-12-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lips Enhancement; Perioral Wrinkles; Nasolabial Fold Wrinkles; Cheek Augmentation; Infraorbital Hollows

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aesthetic treatment with hyaluronic acid (HA) of one or more regions of the face. (Experimental): Based on their preferences and with the agreement of the healthcare professional, subjects may receive aesthetic treatments of the lips, perioral lines, nasolabial folds, cheeks, and/or infraorbital hollows.
  Interventions: Device: Facial injection of hyaluronic acid-based dermal fillers.

INTERVENTIONS:
Device: Facial injection of hyaluronic acid-based dermal fillers. — Facial injection of hyaluronic acid-based dermal fillers USING COLD-X™ TECHNOLOGY by Symatese.

SUMMARY:
The goal of this post-market interventional study is to confirm, under real-life conditions, the safety and performance of hyaluronic acid-based dermal fillers intended to modify skin anatomy and facial appearance. Subjects aged 18 years or older seeking aesthetic treatment of the lips, perioral lines, nasolabial folds, cheeks, and/or infraorbital hollows may be included. The main question the study aims to answer is: How long does the effect of the products last?

Participants will attend follow-up visits every 6 months after the initial injection, until the end of follow-up at 24 months. During each visit, the investigator will assess performance and safety through a simple clinical examination. At each follow-up visit, subjects will also evaluate the aesthetic improvement compared with their pre-injection appearance. Subjects will be asked about the level of pain experienced during the initial injection.

If the subject wishes, a retreatment may be performed at the 12-month or 18-month follow-up visit, provided that the treated area(s) have returned to the pre-injection state.

ELIGIBILITY:
Inclusion Criteria:

* Subject seeking an aesthetic correction of the infraorbital hollows with FASY P and/ or an aesthetic correction of the lips with ESTYME® LIPS, and/ or an aesthetic correction of the perioral lines with ESTYME® SMOOTH, and/ or an aesthetic correction of nasolabial folds with ESTYME® SMOOTH, and/ or an aesthetic correction of cheeks with ESTYME® SCULPT.
* Subject who agreed to participate and have signed an informed consent.
* Age: over 18 years old.
* Subject being affiliated to a health social security system.

Exclusion Criteria:

* Minors
* Subjects with a known allergy to hyaluronic acid, lidocaine or amide local anesthetics.
* Subjects with porphyria.
* Subjects with an autoimmune disorder, or using an immunosuppressant medication.
* Pregnant or breastfeeding women.
* Subjects with inflammation, infection or cutaneous disorders, at the treatment site or nearby.
* Subjects with bleeding disorders or in subjects receiving thrombolytic or anticoagulant treatment.
* Areas other than those recommended by the IFU.
* Subject deprived of liberty by judicial or administrative decision.
* Adults under a legal protection measure (guardianship/curatorship).
* Subject under legal protection order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients returning to their baseline (pre-injection) state for each treated area, based on the investigator's assessment using 5- or 6-point area-specific scales. | At each follow-up visit (6 months, 12 months, 18 months and 24 months)

SECONDARY OUTCOMES:
Injection site reactions (ISR) assessed by the investigators. | D0 (post-first injection), M1 (post optional touch-up), M12/M18 (post optional retreatment)
Number of adverse device effects (ADEs) and serious adverse device effects (SADEs) assessed by the investigators. | From the injection (day 0) to the end of the follow-up period (24 months).
Subject-assessed aesthetic improvement of each treated area, measured using the Global Aesthetic Improvement Scale (GAIS), a 5-point scale ranging from "worse" to "very much improved. | At each visit (Day 0 after injection, day 30 (if any visit), 6 months, 12 months, 18 months and 24 months)
Investigator-assessed aesthetic improvement of each treated area, measured using the Global Aesthetic Improvement Scale (GAIS), a 5-point scale ranging from "worse" to "very much improved. | At each visit (Day 0 after injection, day 30 (if any visit), 6 months, 12 months, 18 months and 24 months)
Investigator-assessed wrinkle severity or volume using 5- or 6-point area-specific scales for each treated area. | At each visit (Day 0 before and after injection, at 30 Days (if any visit), 6 months, 12 months, 18 months, and 24 months)
Subject-reported pain per treated area, rated on an 11-point scale (0 = no pain, 10 = worst pain). | During the initial injection procedure at day 0

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Centre Médical Saint Jean, Arras
  - Cabinet médical, Lyon
  - Palais de Flore, Lyon
  - Centre Laser Palaiseau, Palaiseau
  - Aesthé - Marais., Paris
  - Cabinet médical, Paris
  - Cabinet médical, Saint-Maur-des-Fossés

IPD SHARING:
Plan to Share IPD: No